CLINICAL TRIAL: NCT00085124
Title: A Phase III Study of Daunorubicin and Cytarabine +/- G3139 (Genasense, Oblimersen Sodium, NSC #683428, IND #58842), a BCL2 Antisense Oligodeoxynucleotide, in Previously Untreated Patients With Acute Myeloid Leukemia (AML) > / = 60 Years
Brief Title: Daunorubicin Hydrochloride, Cytarabine and Oblimersen Sodium in Treating Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02805; CALGB-10201; CDR367323; U10CA031946 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities | interventions — oblimersen; Cytarabine; Daunorubicin

ARMS (2):
- Arm I (Experimental): Remission induction therapy: Patients receive oblimersen IV continuously on days 1-10, cytarabine IV continuously on days 4-10, and daunorubicin IV on days 4-6.
  Patients who achieve CR proceed to consolidation therapy. Patients who do not achieve CR receive a second course of induction therapy.
  Second remission induction therapy: Patients receive oblimersen IV continuously on days 1-8, cytarabine IV continuously on days 4-8, and daunorubicin IV on days 4-5.
  Patients who achieve CR proceed to consolidation therapy.
  Consolidation therapy: Patients receive oblimersen IV continuously on days 1-8 and high-dose cytarabine IV over 3 hours on days 4-8. Patients with a continuing CR receive a second course of consolidation therapy.
  Interventions: Biological: oblimersen sodium; Drug: cytarabine; Drug: daunorubicin hydrochloride; Other: laboratory biomarker analysis
- Arm II (Experimental): Remission induction therapy: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV on days 1-3.
  Patients who achieve CR proceed to consolidation therapy. Patients who do not achieve CR receive a second course of induction therapy.
  Second remission induction therapy: Patients receive cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1 and 2.
  Patients who achieve CR proceed to consolidation therapy.
  Consolidation therapy: Patients receive high-dose cytarabine IV over 3 hours on days 1-5. Patients with a continuing CR receive a second course of consolidation therapy.
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
  Arms: Arm I
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial is studying daunorubicin, cytarabine, and oblimersen to see how well they work compared to daunorubicin and cytarabine in treating older patients with previously untreated acute myeloid leukemia. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of daunorubicin and cytarabine by making cancer cells more sensitive to the drugs. It is not yet known whether daunorubicin and cytarabine are more effective with or without oblimersen in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: Primary

I. Compare outcome, in terms of overall survival, disease-free survival, event-free survival, and complete response rate, in older patients with previously untreated acute myeloid leukemia treated with daunorubicin and cytarabine with or without oblimersen.

Secondary I. Determine the significance of expression of select Bcl-2 family member proteins known to be modulated by oblimersen (e.g., Bcl-2) or which potentially mediate resistance to oblimersen (e.g., Bcl-XL or Mcl-1) in predicting clinical outcomes in patients treated with these regimens.

II. Correlate clinical outcomes with serial changes in levels of mRNA and protein expression of Bcl-2, its pro-apoptotic binding partner Bax, and other anti-apoptotic Bax-binding proteins (e.g., Bcl-XL or Mcl-1) in patients treated with these regimens.

III. Determine the effect of pre-treatment characteristics (e.g., morphology, cytogenetics, molecular features, expression of multidrug resistance molecules, functional assays of drug efflux, prior myelodysplastic syndromes, age, and white blood cells) on toxicity of these regimens and outcomes in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I:

Remission induction therapy: Patients receive oblimersen IV continuously on days 1-10, cytarabine IV continuously on days 4-10, and daunorubicin IV on days 4-6.

Patients who achieve complete remission (CR) proceed to consolidation therapy. Patients who do not achieve CR receive a second course of induction therapy.

Second remission induction therapy: Patients receive oblimersen IV continuously on days 1-8, cytarabine IV continuously on days 4-8, and daunorubicin IV on days 4-5.

Patients who achieve CR proceed to consolidation therapy.

Consolidation therapy: Patients receive oblimersen IV continuously on days 1-8 and high-dose cytarabine IV over 3 hours on days 4-8. Patients with a continuing CR receive a second course of consolidation therapy.

Arm II:

Remission induction therapy: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV on days 1-3.

Patients who achieve CR proceed to consolidation therapy. Patients who do not achieve CR receive a second course of induction therapy.

Second remission induction therapy: Patients receive cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1 and 2.

Patients who achieve CR proceed to consolidation therapy.

Consolidation therapy: Patients receive high-dose cytarabine IV over 3 hours on days 1-5. Patients with a continuing CR receive a second course of consolidation therapy.

In both arms, treatment continues in the absence of disease progression, unacceptable toxicity, failure to achieve CR after 2 courses of remission induction therapy, the presence of leukemic cells in the cerebrospinal fluid, leukemic regrowth, or relapse during consolidation therapy.

Patients are followed every 2 months for 2 years, every 3 months for 2 years, and then annually for 10 years.

PROJECTED ACCRUAL: A total of 500 patients (250 per treatment arm) will be accrued for this study within 4.2 years.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE CHARACTERISTICS:

  * Histologically confirmed acute myeloid leukemia
  * No promyelocytic leukemia
  * History of antecedent myelodysplasia allowed provided that the patient received no prior cytotoxic therapy for myelodysplastic syndromes
* PRIOR CONCURRENT THERAPY:

  * Biologic therapy

    * Prior growth factor and/or cytokine support allowed
    * No concurrent routine or prophylactic myeloid growth factors
  * Chemotherapy

    * No prior chemotherapy for leukemia or myelodysplasia except under the following conditions:
    * Emergency leukapheresis
    * Emergency treatment for hyperleukocytosis with hydroxyurea
    * No other concurrent chemotherapy
  * Endocrine therapy

    * No concurrent hormones except steroids for adrenal failure or hormones for non-disease-related conditions allowed (e.g., insulin for diabetes)
  * Radiotherapy

    * Prior cranial radiotherapy for CNS leukostasis (1 dose only) allowed
    * No concurrent palliative radiotherapy
  * Surgery
  * Not specified
  * Other

    * Concurrent enrollment on CALGB-8461, CALGB-9665, and CALGB-9760 allowed
    * No other concurrent investigational or commercial agents or therapies intended to treat the malignancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-12; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 10 years
Complete response (CR) rate | Up to 10 years
Median disease-free survival (DFS) | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Walker AR, Marcucci G, Yin J, Blum W, Stock W, Kohlschmidt J, Mrozek K, Carroll AJ, Eisfeld AK, Wang ES, Jacobson S, Kolitz JE, Thakuri M, Sutamtewagul G, Vij R, Stuart RK, Byrd JC, Bloomfield CD, Stone RM, Larson RA. Phase 3 randomized trial of chemotherapy with or without oblimersen in older AML patients: CALGB 10201 (Alliance). Blood Adv. 2021 Jul 13;5(13):2775-2787. doi: 10.1182/bloodadvances.2021004233. PMID 34251414
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516
- [Derived] Yin J, LaPlant B, Uy GL, Marcucci G, Blum W, Larson RA, Stone RM, Mandrekar SJ. Evaluation of event-free survival as a robust end point in untreated acute myeloid leukemia (Alliance A151614). Blood Adv. 2019 Jun 11;3(11):1714-1721. doi: 10.1182/bloodadvances.2018026112. PMID 31171508
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/